CLINICAL TRIAL: NCT04337047
Title: Distress During the COVID-19 Pandemic in France: a National Assessment of At-risk Populations
Brief Title: Distress in Crisis Situations During COVID-19
Status: Completed | Type: Observational
Sponsor: Wefight (Industry)
Responsible Party: Principal Investigator, benjamin CHAIX, Chief Science Officer, Wefight
Other Study IDs: WefightDistress20
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Vik sein: Vik sein users
  Interventions: Other: questionnaire assesment
- Vik asthme: Vik asthme users
  Interventions: Other: questionnaire assesment
- Vik migraine: Vik migraine users
  Interventions: Other: questionnaire assesment
- Vik depression: Vik depression users
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — questionnaire assesment

SUMMARY:
There are many scales for screening or assessing the impact of a disease. These scales are generally used to diagnose or assess the severity of a disease and are carried out at the request of a physician by the patient. Conversational agents could make it possible to administer these questionnaires remotely, analyse them and use the results on a large scale, without prior medical intervention.

The main objective of this study is to quantify and qualify the distress of a large population in times of pandemic crisis.

DETAILED DESCRIPTION:
The Peritraumatic Distress Inventory is the standard tool designed to assess distress in times of crisis. It consists of 13 questions.

Questions will be submitted to the participants from the Vik chatbot. Responses will be analysed and compared according to the demographics and pathologies encountered.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old

  * Collection of the subject's non-opposition
  * Patient registration on Vik breast, Vik asthma, Vik migraine, Vik depression

Exclusion Criteria:

* Patient unable to formulate non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vik's users in France
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
quantify and qualify distress over a large population in times of pandemic crisis. | 1 month

SECONDARY OUTCOMES:
qualify demographic data vs distress over a large population in times of pandemic crisis. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Wefight, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaix B, Delamon G, Guillemasse A, Brouard B, Bibault JE. Psychological distress during the COVID-19 pandemic in France: a national assessment of at-risk populations. Gen Psychiatr. 2020 Nov 26;33(6):e100349. doi: 10.1136/gpsych-2020-100349. eCollection 2020. PMID 34192239